CLINICAL TRIAL: NCT03426241
Title: The Effect of Smoking on the Expression of Gelatinases in Chronic Periodontitis: A Cross-sectional Study
Brief Title: Effect of Smoking on the Expression of Gelatinases in Chronic Periodontitis
Status: Completed | Type: Observational
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Yasemin Sezgin, Clinician in periodontology department, Baskent University
Other Study IDs: BaskentU2
Record Dates: First submitted 2018-01-29; First posted 2018-02-08 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Periodontitis; Smoking
Keywords: chronic periodontitis; smoking; mmp-2; mmp-9
MeSH Terms: conditions — Periodontitis; Smoking; Chronic Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- smoking chronic periodontitis
  Interventions: Other: no intervention
- non-smoking periodontitis
  Interventions: Other: no intervention
- smoking healthy
  Interventions: Other: no intervention
- non-smoking healthy
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — this is cross-sectional study

SUMMARY:
This study comparatively evaluate the expressions of MMP-2 and MMP-9 in smoker vs non-smoker chronic periodontitis patients as well as periodontally healthy subjects. the hypothesis of this study was that smoking may interfere with periodontal disease by effecting MMP-2 and MMP-9 expressions.

DETAILED DESCRIPTION:
Smokers have greater risk for developing periodontal disease and smoking is highly correlated with greater marginal bone loss. Matrix metalloproteinases (MMP) play a major role in periodontal tissue destruction. MMP-2 and MMP-9, called gelatinases, are one of the major MMPs that plays important roles in periodontitis. To date, several studies showed the increased levels of gelatinases in periodontal disease and only a limited number of study investigated the effect of smoking on gelatinases. However, no previous study has directly investigated the possible relationship between smoking and gingival tissue gelatinases expressions (MMP-2 and MMP-9) in chronic periodontitis (CP) patients relative to periodontally healthy subjects.

Therefore this study is conducted to comparatively evaluate the expressions of MMP-2 and MMP-9 in smoker vs non-smoker chronic periodontitis patients as well as periodontally healthy subjects. the of this study hypothesis was that smoking may interfere with periodontal disease by effecting MMP-2 and MMP-9 expressions.

ELIGIBILITY:
Inclusion Criteria:

* A total of 80 subjects (35 females, 45 males, with an age range of 16-62 years) were included in this study from those patients seeking dental treatment at the Baskent University School of Dentistry between February 2010 and December 2012.

Exclusion Criteria:

* Patients with systemic disease;
* pregnant and/or lactating women;
* patients taking any medications that may influence the study.

Ages: 16 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: A total of 80 subjects (35 females, 45 males, with an age range of 16-62 years) were included in this study from those patients seeking dental treatment at the Baskent University School of Dentistry
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-02-10 (Actual); Primary Completion 2012-12-29 (Actual); Study Completion 2012-12-30 (Actual)

PRIMARY OUTCOMES:
expression of gelatinases levels in gingival tissue among groups | day 1
  In chronic periodontitis group, after recording the clinical parameters, gingival tissues were harvested from the deepest periodontal pocket. Whereas in periodontally healthy group, gingival tissues were collected during crown-lengthening surgery or during an extraction of a teeth for orthodontic reasons. In both groups the samples include both sulcus/pocket epithelium and underlying connective tissues. The expression of MMP-2 and MMP-9 is measured immunohistochemically

SECONDARY OUTCOMES:
difference in probing depths among groups | day o
  Clinical parameters will be recorded and difference in probing depths among the groups will be calculated
difference in probing depths among groups | day 0
  Clinical parameters will be recorded and difference in clinical attahment level among the groups will be calculated

IPD SHARING:
Plan to Share IPD: No